CLINICAL TRIAL: NCT03434236
Title: The Effects of Dietary Supplementation With Lipinova on Inflammatory and Proresolving Lipid Mediator Profiles in Patients Undergoing Total Knee Arthroplasty
Brief Title: The Effects of Lipinova on Inflammatory and Proresolving Lipid Mediator Profiles After Orthopedic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Mieke A. Soens, MD Staff Anesthesiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 2018P000102/PHS
Record Dates: First submitted 2018-02-01; First posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-02

CONDITIONS: Inflammation; Surgery
Keywords: omega-3; specialized proresolving mediators
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Patients will be taking placebo twice daily for 5 days prior to surgery. The placebo has a similar taste and smell as the active supplement.
  Interventions: Dietary Supplement: Placebo
- low dose Lipinova (30mL) (Experimental): Patients will take 15 mL Lipinova (a dietary supplement containing omega-3 PUFA's) twice daily for 5 days prior to surgery.
  Interventions: Dietary Supplement: low dose Lipinova (30 mL daily)
- high dose Lipinova (60mL) (Experimental): Patients will take 30mL of Lipinova (a dietary supplement containing omega-3 PUFA's) twice daily for 5 days prior to surgery.
  Interventions: Dietary Supplement: high dose Lipinova (60mL)

INTERVENTIONS:
Dietary Supplement: low dose Lipinova (30 mL daily) — Lipinova is a nutritional supplement containing concentrated n-3 PUFA (EPA and DHA) and metabolites
  Arms: low dose Lipinova (30mL)
Dietary Supplement: Placebo — Placebo will have a similar appearance, smell and taste as the nutritional supplement
  Arms: Placebo
Dietary Supplement: high dose Lipinova (60mL) — Lipinova is a nutritional supplement containing concentrated n-3 PUFA (EPA and DHA) and metabolites
  Arms: high dose Lipinova (60mL)

SUMMARY:
The aim of this pilot study is to investigate whether pre-operative supplementation with an over the counter dietary supplement containing a fractionated marine lipid concentrate derived from anchovy and sardine oil, Lipinova® (Solutex), improves the inflammatory profile and proresolving capacity in patients undergoing total knee arthroplasty. In addition, the investigators will compare the ability of two different dosing regimens to maximize SPM (Specialized Proresolving Mediators) availability.

DETAILED DESCRIPTION:
The resolution of acute inflammation was once thought to be a passive process, meaning that inflammatory mediators from the acute response (e.g. chemoattractants, complement components, prostaglandins, chemokines and cytokines) would simply dilute and dissipate to stop the infiltration of leucocytes into the tissues. Conversely, more recently it was shown that tissue resolution of inflammation is actually an active programmed process, requiring a temporal lipid mediator class switch that leads to the production of specialized pro-resolving mediators (SPMs) derived from essential fatty acids.1-4

There are several distinct classes of SPMs: the lipoxins derived from the n-6 polyunsaturated fatty acid (n-6 PUFA), AA, and the resolvins, protectins and maresins derived from the n-3 PUFAs, eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA). These SPMs counter regulate pro-inflammatory mediator production, including prostaglandins, leukotrienes, and select cytokines. They also stimulate leucocyte responses including bacterial phagocytosis and efferocytosis of apoptotic cells, key processes in the clearance of infections and return to homeostasis, without apparent immune suppression.5-7 In addition, Serhan and colleagues8 recently identified a new family of sulfido-conjugated mediators that promote wound repair and tissue regeneration. An increasing body of research has shown the beneficial actions of these mediators on improving the inflammatory process in several disease states, such as sepsis, peritonitis, colitis, Alzheimer's disease and peripheral vascular disease.9-13 In addition, it was demonstrated that RvE1 has direct bone-preserving and bone regeneration functions in a mouse model of periodontal disease.14

There is also increasing evidence suggesting that inflammation has a significant impact on postoperative clinical outcomes. Kimura et al.15 demonstrated that patients who developed postoperative infectious complications after liver resection had significantly higher levels of IL-6 on days 0 and 1 after surgery than did those without infections. In addition, elevated pre-operative CRP-levels in patients undergoing palliative surgery is associated with a higher complication rates and decreased overall survival.16 Pillai et al.17 demonstrated two groups among patients undergoing abdominal aorta aneurysm (AAA) surgery based on their temporal profile: one group displayed a pro-inflammatory profile throughout the intra-operative and postoperative time course, while the other group was characterized by a pro-resolving mediator profile. The authors suggested that these two broad categories may reflect an early resolver population and a delayed resolver population and that enhancing the patient profile of endogenous pro-resolving mediators may shorten recovery times, resolution and improve outcomes in these patients.

In this proposal the investigators aim to determine whether pre-operative dietary supplementation with a nutritional supplement containing omega-3 PUFA and its derivatives will improve the metabolo-lipidomic, inflammatory, and resolution profile of patients undergoing total knee arthroplasty. Lipinova® (Solutex) is an over the counter nutritional supplement that differs from other commercially available "Fish Oil" in that it contains standardized levels of the omega 3- PUFAs, Eicosapentaenoic acid (EPA) and Docosahexaenoic acid (DHA) as well as the derived monohydroxylated precursors (17-HDHA, 18-HEPE and 14-HDHA). The standardized levels are obtained from anchovy and sardine oil through advanced fractionation technology and purification technology.

SPECIFIC AIMS:

Specific Aim 1: To characterize the pro-resolving lipid mediator (LM) or specialized pro-resolving mediator (SPM) signature in patients scheduled to undergo total knee arthroplasty. We hypothesize that orthopedic surgery will induce an up-regulation of pro-inflammatory pathways and down-regulation of pro-resolving lipid mediator pathways on postoperative day 1, when compared to pre-operatively.

Specific Aim 2: To determine if pre-operative dietary supplementation with Lipinova®, a purified, fractionated form of fish oil, containing standardized amounts of n-3 essential fatty acids, alters the metabolo-lipidomic profile in patients undergoing total knee arthroplasty. We hypothesize that the oral administration of Lipinova®, which contains precursors for SPMs will upregulate the pro-resolving lipid mediator pathways and down-regulate pro-inflammatory pathways in patients scheduled to undergo total knee arthroplasty, both pre-operatively and on postoperative day 1.

Specific Aim 3: To define a dosing regimen to maximize SPM availability in patients undergoing total knee arthroplasty surgery. We will compare changes in metabolo-lipidomic profiles between patients receiving 2 different doses of Lipinova® supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo total knee arthroplasty at Brigham and Women's Hospital

Exclusion Criteria:

* current treatment with corticosteroids or NSAIDs
* evidence of active infection
* chronic liver disease
* end stage renal disease (CKD-5)
* chronic inflammatory disorders
* recent major illness or surgery within 30 days
* use of immunosuppressive medication
* history of organ transplantation
* pregnancy or plans to become pregnant, or lactating
* allergies to fish or fish oil
* coagulation disorders or thrombocytopenia (platelet < 150,000)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-03-15 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
SPM signature profile/Resolution Index | 6 months
  cumulative levels (in pg/mL) in plasma and serum for DHA-derived SPMs (D-series resolvins: RvD1, RvD2, RvD3, RvD4, RvD5, RvD6, 17R-RvD1 and 17R-RvD3), Protectins (PD1, 17R-PD1), Maresins (MaR1) + EPA-derived SPMs (E-series Resolvins (RvE1, RvE2 and RvE3) + n-3 DPA-derived SPM (RvD1 n-3 DPA, RvD2n-3 DPA and RvD5 n-3 DPA), Protectins (10S, 17S-diHDPA), Marins (MaR1 n-3 DPA) and AA-derived Lipoxins (LXA4, LXB4, 15-epi-LXA4 and 15-epi-LXB4). Cumulative levels (in pg/mL) will be compared before and after treatment with supplement/placebo and before and after surgery. Lipid mediator profiling will be done with LC-MSMS.

CONTACTS AND LOCATIONS:
Overall Officials: Mieke Soens, MD, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: Undecided